CLINICAL TRIAL: NCT01887665
Title: Enhancing Early-Phase Care for Primary Care Patients With Unhealthy Substance Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brandeis University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Elizabeth Merrick, Senior Scientist, Brandeis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12116; 1R21DA032039-01A1 (NIH)
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Substance Use Disorders
Keywords: substance use disorders; substance abuse; substance abuse treatment; contingency management
MeSH Terms: conditions — Substance-Related Disorders | interventions — Fertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Incentives (Experimental): Prize-based financial incentives, informed by contingency management principles, are offered to patients who attend treatment visits.
  Interventions: Behavioral: incentives

INTERVENTIONS:
Behavioral: incentives — A structured system of prize-based financial incentives rewards attendance at treatment visits.

SUMMARY:
The clinical trial portion of this study tests the hypothesis that contingency management-based incentives for primary care patients with substance use disorders to attend treatment services will increase treatment initiation and engagement. The investigators are investigating whether this approach that has been found effective in specialty treatment settings will work in the primary care context, in conjunction with screening.

ELIGIBILITY:
Inclusion Criteria:

* Positive self-report alcohol or drug use screen in primary care
* Diagnosis of substance use disorder
* age 18 or older

Exclusion Criteria:

* SUD treatment in past 60 days
* cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-08; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Initiation | 90 days
  Had initial outpatient treatment visit following positive screen and confirmatory diagnosis
Engagement | 90 days
  Had two additional outpatient treatment visits after initiating treatment

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth L. Merrick, Ph.D., Principal Investigator — Brandeis University
Locations (1):
- Edith Nourse VA Medical Center (Bedford VA), Bedford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No